CLINICAL TRIAL: NCT02967861
Title: Effect of Pranayama on Peroxisome Proliferator-activated Receptor Gamma, Nuclear Factor Kappa B and Red Complex Microorganisms in Patients With Chronic Periodontitis
Brief Title: Effect of Pranayama on Periodontal Health
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Meenakshi Ammal Dental College and Hospital (Other)
Responsible Party: Principal Investigator, Dr.Jaideep Mahendra, Professor, Meenakshi Ammal Dental College and Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAHER-MU-002-IEC/2016
Record Dates: First submitted 2016-11-08; First posted 2016-11-18 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Periodontitis
Keywords: chronic periodontitis; Nuclear factor-kappa B; Pranayama; Peroxisome proliferator - activated receptor gamma; Red complex microorganisms
MeSH Terms: conditions — Chronic Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SRP & pranayama (lifestyle modification) (Active Comparator): 30 chronic periodontitis subjects treated with SRP & pranayama for 3 months
  Interventions: Behavioral: Pranayama
- Scaling and root planing (Placebo Comparator): 30 chronic periodontitis subjects treated with scaling and root planing only
  Interventions: Procedure: Scaling and root planing

INTERVENTIONS:
Behavioral: Pranayama — Pranayama is the breathing exercise through the nostrils. It enhances the systemic immunity which in turn enhances the overall defense mechanism of an individual.
  Arms: SRP & pranayama (lifestyle modification)
Procedure: Scaling and root planing — It is a mechanical debridement of dental plaque.
  Arms: Scaling and root planing

SUMMARY:
The objective of the study was to evaluate the levels of Peroxisome proliferator-activated receptor gamma (PPAR-γ), Nuclear factor-kappa B (NF-kB) and the presence of red complex microorganisms (RCM) such as Treponema denticola (T.d), Porphyromonas gingivalis (P.g) and Tannerella forsythia (T.f) in the subgingival tissues of chronic periodontitis subjects before and after intervention with pranayama as an adjunct to scaling and root planing.

DETAILED DESCRIPTION:
Sixty chronic periodontitis subjects were selected out of which 30 subjects (control group) were treated with scaling and root planing (SRP) and 30 subjects (pranayama group) also underwent SRP and pranayama for 3 months. Clinical parameters were recorded and the presence of PPAR-γ, NF-kB and RCM were assessed at baseline and after 3 months

ELIGIBILITY:
Inclusion Criteria:

* presence of at least 20 teeth
* Probing pocket depth ≥ 5 mm

Exclusion Criteria:

* aggressive periodontitis
* systemic disorders
* pregnant & lactating females
* smokers & alcoholics
* immunocompromised individuals

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy of pranayama in chronic periodontitis patients from baseline to 3 months | 3 months
  Clinical attachment level is measured using Williams periodontal probe in millimeters with the criteria of 1 to 2 mm for slight periodontitis, 3 to 4 mm for moderate periodontits and greater or equal to 5 mm for severe periodontitis.

SECONDARY OUTCOMES:
Microbiological efficacy of pranayama in chronic periodontitis patients from baseline to 3 months | 3 months
  Red complex microorganisms such as P.gingivalis, T.denticola, T.forsythia are identified as '0' for absence and '1' for presence and analysed using polymerase chain reaction from subgingival plaque samples.
Efficacy of pranayama on nuclear factor-kappa B (NF-kB) in chronic periodontitis patients | 3 months
  The expression of NF-kB is analysed using Real time PCR after isolation of RNA from subgingival plaque samples.
Efficacy of pranayama on perosxisome proliferator-activated receptor (PPAR)-γ in chronic periodontitis patients | 3 months
  The expression of PPAR- γ is analysed using Real time PCR after isolation of RNA from subgingival plaque samples.

CONTACTS AND LOCATIONS:
Overall Officials: Jaideep Mahendra, MDS, Ph.D, Principal Investigator — Meenakshi Ammal Dental College & Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Baldwin AS Jr. The NF-kappa B and I kappa B proteins: new discoveries and insights. Annu Rev Immunol. 1996;14:649-83. doi: 10.1146/annurev.immunol.14.1.649. PMID 8717528
- [Result] Pilkington K, Kirkwood G, Rampes H, Richardson J. Yoga for depression: the research evidence. J Affect Disord. 2005 Dec;89(1-3):13-24. doi: 10.1016/j.jad.2005.08.013. Epub 2005 Sep 26. PMID 16185770